CLINICAL TRIAL: NCT06216730
Title: Endoscopic Resection of Papillary Adenomas; a Novel Treatment Algorithm to Prevent Recurrence - a Pilot-study
Acronym: ERASE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERASE- pilot
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Ampullary Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm cohort study (Other): Since this is a single arm cohort study the outcomes will be descriptive
  Interventions: Procedure: Endoscopic papillectomy

INTERVENTIONS:
Procedure: Endoscopic papillectomy — patients undergoing endoscopic papillectomy will be included and treated according to the study algorithm.
  * A papillary adenoma (abnormal tissue growth/ tumour at junction of bile duct & intestines) will be removed completely by cutting & removing abnormal tissue growth using a flexible tube containing a camera through the mouth.
  * After the procedure you will be admitted in the hospital for at least 24 hours for observation,
  * You will be asked to use medications which decrease acid production (PPIs- proton pump inhibitors) in stomach for 2 weeks to decrease the risk of bleeding.

SUMMARY:
Recurrence after endoscopic papillectomy is described in up to 33% of the cases (range 12-33%). This leads to re-interventions, a cumulative risk of adverse events, and the need for long-term follow-up. Recurrences most likely originate from either the biliary orifice or lateral resection margins. Ablative methods such as radiofrequency ablation (RFA) and thermal ablation by cystotome inside the bile duct have been described to treat intraductal extension of which the use of a cystotome seems to have a more favorable safety profile. However, no studies focusing on the preventive use of these ablative methods in patient with papillary adenomas have been performed.

DETAILED DESCRIPTION:
Recurrence after endoscopic papillectomy is described in up to 33% of the cases (range 12-33%). This leads to re-interventions, a cumulative risk of adverse events, and the need for long-term follow-up. Recurrences most likely originate from either the biliary orifice or lateral resection margins. Ablative methods such as radiofrequency ablation (RFA) and thermal ablation by cystotome inside the bile duct have been described to treat intraductal extension of which the use of a cystotome seems to have a more favorable safety profile. However, no studies focusing on the preventive use of these ablative methods in patient with papillary adenomas have been performed. It is hypothesized that the curative resection rate can be increased and recurrence prevented by using a combination of snare tip soft coagulation (STSC) of the resection margins and thermal ablation by cystotome of the biliary orifice in patients with and without the suggestion of intraductal extension

ELIGIBILITY:
Inclusion Criteria:

* Papillary adenoma which seems suitable for curative endoscopic resection.
* 18 years or older.
* Capable of providing written and oral informed consent.

Exclusion Criteria:

* Patients with intraductal extension of >1 cm beyond the duodenal wall or adenocarcinoma will be excluded since surgical resection is considered the preferred treatment in these cases.(16)
* Failure to place a PD stent in patients with normal pancreatic duct anatomy.
* Refusal to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-05 (Estimated); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Primary outcome will be safety i.e. rate of adverse events such as pancreatitis, bleeding, cholangitis, perforation, and papillary stenosis (at 9 months follow-up). | 1 YEAR(2024-2025)
  rate of adverse events such as pancreatitis, bleeding, cholangitis, perforation, and papillary stenosis (at 9 months follow-up).

IPD SHARING:
Plan to Share IPD: No